CLINICAL TRIAL: NCT06029452
Title: A Retrospective Chart Validation Study Evaluating the Performance of Machine Learning Algorithm (ML) to Predict the Clinical Diagnosis of Wild-type Transthyretin Amyloid Cardiomyopathy (ATTRwt-CM) and Non-amyloid Heart Failure Among Patients With Heart Failure (HF)
Brief Title: A Retrospective Validation Study To Identify Chart-Based Clinical Diagnosis Of Wild-Type Transthyretin Amyloid Cardiomyopathy (Attrwt-CM) And Non-Amyloid Heart Failure Among Patients With Heart Failure (HF).
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B3461111
Record Dates: First submitted 2023-09-01; First posted 2023-09-08 (Actual); Results first posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-11

CONDITIONS: ATTR-CM
Keywords: Chronic Heart Failure
MeSH Terms: interventions — Machine Learning Algorithms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- ATTRwt-CM and non-amyloid heart failure patients
  Interventions: Other: Machine learning algorithm

INTERVENTIONS:
Other: Machine learning algorithm — Software to calculate the predicted probability of ATTRwt-CM for these heart failure patients based on the presence and absence of certain features

SUMMARY:
This is an observational, retrospective non-inferiority study with a study sample from a large national database.

A machine learning (ML) model will use a national database to predict the clinical diagnosis of ATTRwt-CM among HF patients. This study will include HF patients ≥50 years old.

ELIGIBILITY:
Inclusion Criteria:

* HF patients (defined as having ≥1 claim for HF or HF treatment) ≥50 years old with clinical diagnosis of ATTRwt-CM or non-amyloid HF ascertained by charts. Patients will be required to have ≥12 months of continuous activity in the EHR or claims prior to the Index Date.

Exclusion Criteria:

* Patients with any of the following diagnoses:

  * Light chain (AL) amyloidosis
  * Intracranial hemorrhage
  * Cerebral amyloid angiopathy
  * End stage renal disease
  * Blood cancer

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart failure patients with clinical diagnosis of ATTRwt-CM or non-amyloid HF
Sampling Method: Non-Probability Sample
Enrollment: 558 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-11-14 (Actual); Study Completion 2023-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B3461111

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with heart failure (HF) who met the inclusion and exclusion criteria were identified from the Optum electronic healthcare records (EHR) database between 01 January 2018 & 30 April 2023 (approximately 5.4 years). Participants with clinical diagnosis of wild-type transthyretin amyloid cardiomyopathy (ATTRwt-CM) or non-amyloid HF were included in this retrospective study chart validation study. Available data was evaluated from 01 September 2023 to 14 November 2023 (up to 2.5 months).
Groups:
- ATTRwt-CM Participants: Participants with clinical diagnosis of ATTRwt-CM between 01 January 2018 to 30 April 2023 were observed in this retrospective study. Available data of eligible participants were studied for 2.5 months in this retrospective observational study.
- Non-amyloid HF Participants: Participants with clinical diagnosis of non-amyloid HF between 01 January 2018 to 30 April 2023 were observed in this retrospective study. Available data of eligible participants were studied for 2.5 months in this retrospective observational study.
Period: Overall Study
Arm/Group | ATTRwt-CM Participants | Non-amyloid HF Participants
Started | 238 | 320
Completed | 238 | 320
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study population included all eligible participants with clinical diagnosis of ATTRwt-CM and Non-amyloid HF whose data was retrieved and evaluated in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | ATTRwt-CM Participants | Non-amyloid HF Participants | Total
Number analyzed (Participants) | 238 | 320 | 558
Age, Customized [Count of Participants; unit: Participants]
  50 to 65 Years | 11 | 73 | 84
  >=65 years | 227 | 247 | 474
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 238 | 320 | 558
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants According to Clinical Diagnosis Predicted Using the Machine Learning (ML) Algorithm
Description: In this outcome measure number of participants were reported according to clinical diagnosis predicted by ML algorithm. True positive (TP) = participants with actual and predicted diagnosis of ATTRwt-CM; False positive (FP) = participants with actual diagnosis of non-amyloid HF and predicted diagnosis of ATTRwt-CM; False negative (FN) = participants with actual diagnosis of ATTRwt-CM and predicted diagnosis of non-amyloid HF; True negative (TN) = participants with actual and predicted diagnosis of non-amyloid HF.
Time Frame: At diagnosis, anytime during retrospective data identification period of approximately 5.4 years; retrospective data observed in this study for approximately 2.5 months
Population: Study population included all eligible participants with clinical diagnosis of ATTRwt-CM and Non-amyloid HF whose data was retrieved and evaluated in the study. Here, "Number of Participants Analyzed" signifies number of participants with respective actual clinical diagnosis ascertained by medical charts.
Measure: Count of Participants; unit: Participants
Arm/Group | ATTRwt-CM Participants | Non-amyloid HF Participants
Number analyzed (Participants) | 238 | 320
Participants
  Predicted for ATTRwt-CM | 203 | 133
  Predicted for Non-amyloid HF | 35 | 187
Statistical Analysis 1: Comparison: ATTRwt-CM Participants vs Non-amyloid HF Participants; Test type: Non-Inferiority — Non-inferiority margin was 0.10; Sensitivity = 0.853, 95% CI 1-sided [lower limit 0.815] — Sensitivity was defined as the probability that an individual with the disease in the population were screen positive for disease by the algorithm (TP). Sensitivity = TP / (TP + FN)
Statistical Analysis 2: Comparison: ATTRwt-CM Participants vs Non-amyloid HF Participants; Test type: Non-Inferiority — Non-inferiority margin was 0.10; Specificity = 0.584, 95% CI 1-sided [lower limit 0.539] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Not applicable as adverse events were not collected for the study
Description: Due to non-interventional nature of study and nature of data sources, the minimum criteria for reporting an adverse event (that is, identifiable participant, identifiable reporter, a suspect product, and event) could not be met, hence adverse events were not planned to be collected and reported.
Arm/Group | ATTRwt-CM Participants | Non-amyloid HF Participants
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-27): https://cdn.clinicaltrials.gov/large-docs/52/NCT06029452/Prot_SAP_000.pdf